CLINICAL TRIAL: NCT00617760
Title: Open-label, Randomized, 3-arm, Phase 3B Clinical Study to Investigate the Safety and Immunogenicity of a Concomitant Administration of Group C Meningococcal Polysaccharide-Tetanus Toxoid Conjugate (MenC-TT) Vaccine and 7-valent Pneumococcal CRM197-conjugate Vaccine (PCV7) in Toddlers Previously Immunized During Infancy With PCV7
Brief Title: Safety and Immunogenicity Study of MenC-TT Vaccine (NeisVac-C) in Toddlers Previously Immunized With PCV7 (Prevenar®)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 670701
Record Dates: First submitted 2008-02-06; First posted 2008-02-18 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Neisseria Meningitidis (Bacterial Meningitis); Invasive Pneumococcal Disease (IPD)
MeSH Terms: conditions — Meningitis, Bacterial | interventions — Vaccines; Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Concomitant administration of MenC-TT vaccine and PCV7, 170 subjects
  Interventions: Biological: Group C Meningococcal Polysaccharide-Tetansu Toxoid Conjugate (MenC-TT) vaccine and 7-valent Pneumococcal CRM197-conjugate vaccine (PCV7)
- 2 (Active Comparator): PCV7 administration only, 85 subjects
  Interventions: Biological: 7-valent Pneumococcal CRM197-conjugate vaccine (PCV7)
- 3 (Active Comparator): MenC-TT vaccine only, 85 subjects
  Interventions: Biological: Group C Meningococcal Polysaccharide-Tetansu Toxoid Conjugate (MenC-TT)

INTERVENTIONS:
Biological: Group C Meningococcal Polysaccharide-Tetansu Toxoid Conjugate (MenC-TT) vaccine and 7-valent Pneumococcal CRM197-conjugate vaccine (PCV7) — MenC-TT vaccine (0.5 ml) to be administered in the left thigh muscle, PCV7 (0.5 ml) to be administered in the right thigh muscle
  Other Names: NeisVac-C and Prevenar®
  Arms: 1
Biological: 7-valent Pneumococcal CRM197-conjugate vaccine (PCV7) — PCV7 (0.5 ml) to be administered in the right thigh muscle
  Other Names: Prevenar®
  Arms: 2
Biological: Group C Meningococcal Polysaccharide-Tetansu Toxoid Conjugate (MenC-TT) — MenC-TT vaccine (0.5 ml) to be administered in the left thigh muscle
  Other Names: NeisVac-C
  Arms: 3

SUMMARY:
The purpose of this study in healthy toddlers who have not previously been immunized against MenC infection and who completed their primary immunization series with PCV-7 (3 vaccinations) during infancy is to demonstrate that the concomitant administration of a single dose of MenC-TT vaccine and a PCV7 booster does not influence the immune response to the seven pneumococcal strains contained in PCV7 as compared to administration of PCV7 alone, and does not influence the immune response to the MenC-TT vaccine as compared to administration of MenC-TT vaccine alone.

ELIGIBILITY:
Inclusion Criteria:

Male and female subjects will be eligible for participation in this study if:

* they are toddlers, aged 12 to 18 months
* they are clinically healthy (i.e. the physician would have no reservations vaccinating with a MenC conjugate vaccine, and/or PCV7 outside the scope of a clinical trial)
* their parents/legal guardian(s) understand the nature of the study, agree to its provisions, and provide written informed consent
* their parents/legal guardian(s) agree to keep a Subject Diary
* they have received a complete primary series of pneumococcal conjugate vaccine (3 vaccinations with PCV7 in the first year of life according to the official vaccination calendar recommendations)

Exclusion Criteria:

Subjects will be excluded from participation in this study if:

* they have a history of any vaccine-related contraindicating event, e.g. serious reactions after first application of a PCV7 vaccine or high fever >= 40ºC associated with any vaccination, or generalized allergic reaction within 48 hours of a first application of vaccine
* they have a known sensitivity or allergy to any components of the vaccines
* they have previously been vaccinated with MenC vaccine
* they have already received a PCV 7 booster (4th vaccination)
* they have a rash or other dermatological condition at the injection site which could interfere with injection site reaction evaluation
* they suffer from a disease (e.g. autoimmune disease) or are undergoing a form of treatment (e.g. systemic corticosteroids) that can be expected to influence immunological functions
* they have a history of meningococcal serogroup C and/or invasive pneumococcal infection
* they have received any blood products or immunoglobulins within 90 days of study entry or the administration of such products is planned during the study period
* currently have or had a history of any serious disease (e.g. cardiac, renal, autoimmune, neurologic)
* were administered an investigational drug within 6 weeks prior to study entry or are concurrently participating in a clinical study that includes the administration of an investigational product
* they or their parents /legal guardian(s) are in a dependent relationships with the study investigator or with a study team member. Dependent relationships include close relatives (i.e., children or grandchildren, partner/spouse, siblings) as well as employees of the investigator or site conducting the study.

Ages: 12 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 330 (Actual)
Dates: Start 2008-03; Primary Completion 2009-08 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Number of subjects achieving PCV7-specific (elicited by each vaccine pneumococcal serotype) antibody concentrations of at least 0.2 mg/mL 1 month after a booster vaccination with PCV7 | 1 month after booster vaccination with PCV7
Number of subjects achieving sero-protective levels of meningococcal serogroup C (MenC) specific serum bactericidal activity (SBA), defined as titer >=1:8, 1 month after administration of MenC-TT vaccine | 1 month after administration of MenC-TT vaccine

CONTACTS AND LOCATIONS:
Locations (27):
- Germany (27):
  - Werderstrasse 3, Bad Saulgau, Baden-Wurttemberg
  - Hauptstrasse 9, Bietigheim-Bissingen, Baden-Wurttemberg
  - Kirchstrasse 2, Bönnigheim, Baden-Wurttemberg
  - Winckelhoferstrasse 3, Ehingen, Baden-Wurttemberg
  - Rheinstrasse 13, Ettenheim, Baden-Wurttemberg
  - Hauptstrasse 240, Kehl, Baden-Wurttemberg
  - Schwarzwaldstrasse 20, Kirchzarten, Baden-Wurttemberg
  - Bismarkstrasse 3, Ludwigsburg, Baden-Wurttemberg
  - Flattichstrasse 29, Ludwigsburg, Baden-Wurttemberg
  - Wilhelmstrasse 25, Metzingen, Baden-Wurttemberg
  - Grossbottwarer Strasse 47, Oberestenfeld, Baden-Wurttemberg
  - Bergstrasse 27, Rottweil, Baden-Wurttemberg
  - Königstrasse 35, Rottweil, Baden-Wurttemberg
  - Crailsheimer Strasse 63, Schwäbisch Hall, Baden-Wurttemberg
  - Schillerstrasse 11, Tuttlinger, Baden-Wurttemberg
  - Broner Platz 6, Weingarten, Baden-Wurttemberg
  - Neuschwansteinstrasse 5, Augsburg, Bayern (Bavaria)
  - Lehenstrasse 12, Bindlach, Bayern (Bavaria)
  - Mohrenstrasse 8, Coburg, Bayern (Bavaria)
  - Bahnhofstrasse 13, Ebersberg, Bayern (Bavaria)
  - Löpsingerstrasse 8, Nördlingen, Bayern (Bavaria)
  - Falkensteiner Strasse 24, Roding, Bayern (Bavaria)
  - Langenbeckstrasse 1, Mainz, Rhineland-Palatinate
  - Goethestrasse 30, Arnstadt, Thuringia
  - Schloß-Prunn-Str. 1, Munich
  - Schwarzwaldstr. 18, Oberkirch
  - Christofstr.13A, Schwieberdingen